CLINICAL TRIAL: NCT00611611
Title: BLyS and IFN Responses to Antigen Challenge in Human SLE
Brief Title: BLYS and IFN in SLE
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Hospital for Special Surgery, New York (Other)
Responsible Party: W Winn Chatham, University of Alabama at Birmingham
Other Study IDs: F060217005; NIH R21 AI069363
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Influenza Vaccines; Pneumococcal Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: SLE
  Interventions: Biological: fluzone; Biological: pneumovax
- 2: healthy controls
  Interventions: Biological: fluzone; Biological: pneumovax

INTERVENTIONS:
Biological: fluzone — once
Biological: pneumovax — once

SUMMARY:
This protocol tests whether changes in BLyS or IFN can be detected in a normal immune response to a vaccine and, if so, whether the response differs between those with lupus and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* ACR lupus criteria
* 18<age<65

Exclusion Criteria:

* chronic infection or cancer
* pregnancy

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: lupus and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
change in specific antibodies in response to vaccine | 2 weeks

SECONDARY OUTCOMES:
change in BLyS after vaccination | 2 weeks
change in IFN after vaccination | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Carter, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States